CLINICAL TRIAL: NCT02910843
Title: Neoadjuvant Treatment With Regorafenib and Capecitabine Combined With Radiotherapy in Locally Advanced Rectal Cancer. A Multicenter Phase Ib Trial (RECAP)
Brief Title: Neoadjuvant Treatment With Regorafenib and Capecitabine Combined With Radiotherapy in Locally Advanced Rectal Cancer
Acronym: RECAP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to structural financial deficit of SAKK
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/16 - RECAP
Record Dates: First submitted 2016-09-14; First posted 2016-09-22 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; Neoadjuvant treatment; Regorafenib; Capecitabine; locally advanced rectal cancer; Phase Ib trial
MeSH Terms: conditions — Rectal Neoplasms | interventions — regorafenib; Capecitabine; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib & Capecitabine (Experimental): * Regorafenib dose level 1-3: day 1 to 14 and day 22 to 35 (2 weeks on 1 week off, 2 weeks on, including Saturday and Sunday) at a daily dose according to the escalation table.
  * Regorafenib dose level -1: day 1 to 5, day 8 to 12, day 22 to 26 and day 29 to 33 (5 days on and 2 days off during week 1, 2, 4 and 5; week 3 off) at a daily dose according to the escalation table.
  * Capecitabine: day 1 to 38 (5 weeks and 3 days, including Saturday and Sunday) according to dose escalation table. The intake stops in the evening of the last day of RT.
  * External beam Radiotherapy
  * Surgery
  Interventions: Drug: Regorafenib; Drug: Capecitabine; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Regorafenib — * Regorafenib dosel level 1-3: day 1 to 14 and day 22 to 35 (2 weeks on 1 week off, 2 weeks on, including Saturday and Sunday) at a daily dose according to the escalation table.
  * Regorafenib dosel level -1: day 1 to 5, day 8 to 12, day 22 to 26 and day 29 to 33 (5 days on and 2 days off during week 1, 2, 4 and 5; week 3 off) at a daily dose according to the escalation table.
  Other Names: BAY 73-4506
Drug: Capecitabine — • Capecitabine: day 1 to 38 (5 weeks and 3 days, including Saturday and Sunday) according to dose escalation table. The intake stops in the evening of the last day of RT.
  Other Names: XELODA
Radiation: Radiotherapy — Monday through Friday for 5 weeks and 3 days (d1-38) starting on day 1 (daily fraction 1.8 Gy, final dose 50.4 Gy).
Procedure: Surgery — 6-12 weeks (± 1 week) after radio-chemotherapy (RCT) has been completed (42-84 days after last day of RCT).

SUMMARY:
Despite treatment of locally advanced rectal cancer relapses are frequent. Several attempts to improve these results with therapy intensification have shown modest effect on disease free survival (DFS) and overall survival (OS). Recent studies with addition of sorafenib and cediranib revealed promising effect on tumor response with acceptable toxicity. Regorafenib is a multi tyrosine kinase inhibitor (TKI) with a broad mechanism of action. Therefore this trial investigates if similar results can be achieved as with sorafenib or cediranib.

DETAILED DESCRIPTION:
Despite treatment of locally advanced rectal cancer relapses are frequent. Several attempts to improve these results with therapy intensification have shown modest effect on disease free survival (DFS) and overall survival (OS). Recent studies with addition of sorafenib and cediranib revealed promising effect on tumor response with acceptable toxicity. Regorafenib is a multi tyrosine kinase inhibitor (TKI) with a broad mechanism of action. Therefore this trial investigates if similar results can be achieved as with sorafenib or cediranib.

The objective of the dose escalation part is to determinate safety, tolerability and the recommended dose. The objective of the expansion cohort is to assess the efficacy and to further characterize safety and tolerability of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before any trial specific procedures.
* Histologically confirmed and clinically advanced adenocarcinoma. pStage 2 and 3 according AJCC 2012, mrT3/4 N0, mrTx N1-2 cM0 (assessed by mandatory CT scan thorax/abdomen, MRI pelvis). TNM classification; recommended MRI quality assurance.
* Tumor is located in the lower and middle rectum (caudal end is defined at maximum of 12 cm from anal verge measured by endoscopy).
* A multi-disciplinary tumor board recommends neoadjuvant radio-chemotherapy and surgery.
* No DPD deficiency (Dihydro-pyrimidine-dehydrogenase DPD deficiency test mandatory). Carrier status of a predefined risk allele of the dihydro-pyrimidine-dehydrogenase gene (DPYD), defined as the presence of at least one of the following mutations: c.1679T>G, c.1905+1G>A, c.2846A>T, c.1129-5923C>G.
* Age 18 to 75 years.
* WHO performance status 0-1.
* Adequate bone marrow function: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 100 g/L.
* Adequate hepatic and pancreatic function: bilirubin ≤ 1.5 x ULN, AST/ALT/AP ≤ 2.5 x ULN, Lipase ≤ 1.5 x the ULN.
* Adequate renal function (calculated creatinine clearance > 50 mL/min, according to the formula of Cockcroft-Gault).
* INR ≤ 1.5 or PTT ≤ 1.5 x ULN (patients who are being therapeutically anticoagulated are not allowed to participate in the trial). If anti coagulation is indicated during trial treatment, low molecular weight heparin must be used.
* Women with child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant during trial treatment and during the 8 weeks thereafter. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential.
* Men agree to use effective contraception during trial treatment and 8 weeks thereafter.

Exclusion Criteria:

* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Concurrent or recent (within 30 days of registration) treatment with any other experimental drug.
* Any prior treatment for rectal cancer.
* Major surgery or significant traumatic injury within 28 days before registration (colostomy accepted).
* Concomitant strong CYP3A4 inhibitors (e.g. clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (e.g. carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort) within 28 days or 5 drug half-lives (if drug half-life in patients is known), whichever is shorter, before start of trial treatment (see http://medicine.iupui.edu/).
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA II-IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation (QTc interval >460 msec), uncontrolled hypertension (sustained systolic blood pressure > 150 mm Hg and/or diastolic > 100 mm Hg despite antihypertensive therapy).
* Patients with evidence or history of any bleeding diathesis, irrespective of severity.
* Any hemorrhage or bleeding event ≥ Grade 3, NCI-CTCAE v4.03 within 4 weeks prior to the start of trial medication.
* Significant proteinuria: Positive dipstick 2+ and greater if proteinuria ≥ 3.5g/24 h measured by urine protein-creatinine ratio is confirmed (≥ Grade 3, NCI-CTCAE v4.0).
* Patients with known hepatopathy as cirrhosis or diseases like Morbus Gilbert Meulengracht.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* History of organ allografts.
* Known hypersensitivity to any of the trial drugs, trial drug classes, or excipients in the formulation.
* Breast-feeding patients.
* Any concomitant drugs contraindicated for use with the trial drugs according to the Swissmedic approved product information.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLTs) | up to 4 weeks after the last administration of RCT
  In the dose escalation part the dose limiting toxicity (DLTs) is observed during and up to 4 weeks after the last administration of RCT.
Pathological near complete or complete tumor response (npCR or pCR) | up to 2 months after end of treatment
  In the dose escalation part the pathological near complete or complete tumor response (npCR or pCR) is specified.

SECONDARY OUTCOMES:
Quality of the mesorectal excision including details of the circumferential resection margin (CRM)/surface | up to 2 months after end of treatment
  Quality of the mesorectal excision including details of the circumferential resection margin (CRM)/surface according to Nagtegaal.
Sphincter preservation | up to 2 months after end of treatment
  Sphincter preservation is defined as preservation of the rectal sphincter or part of it.
Pathological response | up to 2 months after end of treatment
  Dworak tumor regression grading (TRG) system.
Circumferential resection margin (CRM) status | up to 2 months after end of treatment
  Negative (clear) circumferential margins are defined by an invasion front which is at a > 1mm distance from the lateral resection margin; circumferential resection margins of ≤ 1 mm are considered positive (involved).
  CRM negative (clear) ≤ 1mm and CRM positive (involved) ≤ 1mm.
Downstaging of primary tumor and/or lymph nodes (comparison between mrT/N and ypT/N) | up to 2 months after end of treatment
  Downstaging of primary tumor and/or lymph nodes (comparison between mrT/N and ypT/N)
Postoperative complications | within 8 weeks after surgery
  Surgical complications within 8 weeks after surgery. A surgical local complication is defined as either:
  * insufficiency of anastomosis
  * fistula
  * severe local infection requiring antibiotics
  * bladder dysfunction
  * erectile dysfunction
  * additional interventions / operation needed (e.g. drainage of hematoma/abscess)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bastian, MD, Study Chair — Kantonsspital Graubünden, Chur
Locations (7):
- Switzerland (7):
  - St. Claraspital Basel, Basel
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No